CLINICAL TRIAL: NCT06176430
Title: Comparison of Twice Weekly Versus Daily Iron Therapy in Treating Anemia in Children With Cerebral Palsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Dr Yusra Kafait, Pediatrics Resident, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F.1-1/2015/ERB/SZABMU/747
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy; Iron Deficiency Anemia
Keywords: cerebral palsy, anemia
MeSH Terms: conditions — Cerebral Palsy; Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: laboratory personnel only will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily Group (Active Comparator): one group will receive ferrous sulphate 3mg/kg in the form of syrup daily
  Interventions: Drug: Ferrous Sulfate Oral Product
- Twice Weekly Group (Sham Comparator): other group will receive ferrous sulphate 3mg/kg in the form of syrup twice weekly.
  Interventions: Drug: Ferrous Sulfate Oral Product

INTERVENTIONS:
Drug: Ferrous Sulfate Oral Product — ferrous sulphate oral in the form of syrup

SUMMARY:
a randomized clinical trial to compare the effect of twice weekly versus daily iron therapy in treating anemia in children with cerebral palsy, to be conducted at Department of pediatric medicine children's hospital PIMS islamabad.

DETAILED DESCRIPTION:
a total of 160 children of either gender with age between 6 and 60 months diagnosed with cerebral palsy and concomitant iron deficiency anemia will be enrolled, they will be allocated two groups by lottery method. one group will be given ferrous sulphate 3mg/kg daily in the form of syrup and other group will be given ferrous sulphate 3mg/kg twice weekly in the form of syrup for a period of 4 weeks. the primary outcome will be measured as rise in hemoglobin levels more than or equal to 1g/dl at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All the children with cerebral palsy who are diagnosed cases of iron deficiency anaemia
2. Age 06 months to 5 years
3. Both genders

Exclusion Criteria:

1. >5 years of age
2. Children with severe anaemia requiring transfusion (Hb<5 g/L)
3. Children with history of taking oral/IV iron supplements or repeated blood transfusions during last one month
4. Children with concomitant diarrheal disease
5. Where parents are not willing to participate in the study

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin levels from baseline | 4 weeks
  rise in Hb at the end of 4 weeks as more than equal to 1g/dl

SECONDARY OUTCOMES:
Mean change in MCV (Mean Corpuscular Volume) | 4 weeks
  mean change from baseline at the end of 4 weeks
Mean change in mean corpuscular hemoglobin concentration (MCHC) | 4 weeks
  mean change from baseline at the end of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yusra Kafait, MBBS, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University